CLINICAL TRIAL: NCT06739577
Title: Show Me How You Move and I Will Tell You Who You Are. Body Movement Analysis and Automatic Recognition of Associated Vestibular Impairment Patterns
Brief Title: Show Me How You Move and I Will Tell You Who You Are
Status: Completed | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: ABMA
Record Dates: First submitted 2024-12-10; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Vestibular Disease; Vestibular Function Disorder
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Vestibular: Patients with vestibular loss diagnosed by senior ENT doctors with the gold standard ENT measures (caloric testing, head impulse test and/or vestibular evoked myogenic potential, ocular and cervical)
  Interventions: Diagnostic Test: Evaluation of walking abilities (manual Timed-Up & Go - TUG and automatic -OpenTUG)); Diagnostic Test: Neuropsychological assesment is provide to measure objective and subjective cognition/emotional aspects.
- Healthy controls: People with no vestibular loss
  Interventions: Diagnostic Test: Evaluation of walking abilities (manual Timed-Up & Go - TUG and automatic -OpenTUG)); Diagnostic Test: Neuropsychological assesment is provide to measure objective and subjective cognition/emotional aspects.

INTERVENTIONS:
Diagnostic Test: Evaluation of walking abilities (manual Timed-Up & Go - TUG and automatic -OpenTUG)) — To evaluate walking abilities, participants performed the Timed-Up & Go (TUG) f our times (practice trial, normal, slow and fast speed). Patient's performances are videorecorded with an Intel RealSense depth camera D435i to capture their movements, and manual time recording of time taken (in seconds) and number of steps are carried out by the experimenters.
  Complementary to manual experimenter recording, a 2D human pose estimation method (OpenTUG) is applied to automatically extract the time and the number of steps taken by the participant during the TUG task.
  Other Names: Neuropsychological assesment
Diagnostic Test: Neuropsychological assesment is provide to measure objective and subjective cognition/emotional aspects. — Neuropsychological evaluation assess attention (Test for Attentional Performance -TAP-) and quality-of-life (DHI, HADS, and NVI).

SUMMARY:
The aim of this experiment is to gain a better understanding of the body movement patterns of patients with balance disorders (following damage to the vestibular system), as well as their cognitive performance profile. To achieve this, we will need to assess the performance of both patients and healthy subjects with no balance disorders. We will be using a newly-developed artificial intelligence tool to analyze body movement patterns on the basis of participants' videos, and we will also be evaluating participants' performance in a few simple tests of reaction times to image presentations on computer and/or tablet/smartphone.

If you agree to take part in this experiment, you will be asked to perform a simple walking exercise in a corridor (filmed and supervised by a physiotherapist) as well as a few objective cognitive measurement tests (reaction time to attentional and vigilance tasks on computer and/or tablet/smartphone) and subjective tests (self-reported questionnaires) requiring around 40 minutes of investigation in total.

In the long term, the results of this research will make it easier to assess balance disorders in patients with vestibular pathology, and better quantify any cognitive difficulties they may have.

ELIGIBILITY:
For patients :

Inclusion Criteria:

* Age between 18 and 90 years old.
* Vestibular loss diagnosed by senior ENT doctors with the gold standard ENT measures (caloric testing, head impulse test and/or vestibular evoked myogenic potential, ocular and cervical).

Exclusion Criteria:

* Previous neurological disorders (stroke, dementia, …)
* Current medication interfering with the testing (reducing reaction time).
* Visual difficulties interfering with the testing (Visual field reduction,…)
* Age below 18 years old.

For healthy controls :

Inclusion criteria :

- Age between 18 and 90 years old.

Exclusion criteria:

* Previous neurological disorders (stroke, dementia, …)
* Current medication interfering with the testing (reducing reaction time)
* Visual difficulties interfering with the testing (Visual field reduction,…)
* Vertigo or balance complains or an history of previous vestibular disorder.
* Age below 18 years old.
* Not being able to understand the consigns of the task.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Vestibular loss diagnosed by senior ENT doctors with the gold standard ENT measures (caloric testing, head impulse test and/or vestibular evoked myogenic potential, ocular and cervical).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Neuropsychological measures | Through the entire study, approximately 24 months
  evaluation to assess attention (Test for Attentional Performance -TAP-) Alertness and Divided attention tasks. Median reaction time and standard deviation of the median (regularity) are record in milliseconds. Slow reaction times and large standard deviations indicate more difficulties.
Neuropsychological measures | Through the entire study, approximately 24 months
  evaluation to assess quality-of-life (DHI -Dizziness Handicap Inventory, Jacobson & Newman, 1990, Demanez 1991) 25-items, each scored on a 5-point Likert scale. Covering three main areas of difficulties: functional, physical, and emotional aspects related to dizziness and instability.
  Higher scores = higher complains
Neuropsychological measures | Through the entire study, approximately 24 months
  evaluation to assess quality-of-life (Anxiety and depression symptoms, measured with the French version of the Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983), using a 14-item self-assessed questionnaire, each with a 4-point response Likert scale.
  Higher scores = higher complains
Neuropsychological measures | Through the entire study, approximately 24 months
  evaluation to assess subjective perception of cognitive difficulties associated to vertigo with the Neuropsychological Vertigo Inventory - NVI (Lacroix et al., 2016), using 28-items, each scored on a 5-point Likert scale and divided into 7 distinct subscales measuring attention, memory, emotion, space perception, time perception, vision, and motor abilities.
  Higher scores = higher complains
Walking activity | Through the entire study, approximately 24 months
  Participants performed the Timed-Up & Go (TUG) four times (practice trial, normal, slow and fast speed). They have to stand up from a chair, walk until a line on the ground marked at 3 meters, turn, go back to the chair, and sit down again. The time is recorded. There is no time limit to the task.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No